CLINICAL TRIAL: NCT01111773
Title: An Open-label Pilot Study Evaluating Synera® in the Treatment of Patients With Patellar Tendinopathy
Brief Title: Study Evaluating a Heated Lidocaine and Tetracaine Topical Patch in the Treatment of Patients With Patellar Tendinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-204
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Patellar Tendinopathy
Keywords: Patellar tendonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heated Lidocaine and Tetracaine Patch (Experimental)
  Interventions: Drug: Heated Lidocaine and Tetracaine Patch

INTERVENTIONS:
Drug: Heated Lidocaine and Tetracaine Patch — Patients will apply one lidocaine 70 mg and tetracaine 70 mg topical patch to the affected knee twice daily for approximately 14 days. Patches will be applied morning and evening (applications separated by approximately 8-10 hours).
  Other Names: Synera

SUMMARY:
The purpose of the study is to explore the potential usefulness of a heated lidocaine 70 mg and tetracaine 70 mg topical patch for the treatment of pain associated with patellar tendinopathy.

DETAILED DESCRIPTION:
The purpose of this pilot study is to explore the potential usefulness of a heated lidocaine 70 mg and tetracaine 70 mg topical patch for the treatment of pain associated with patellar tendinopathy. A number of efficacy variables will be employed to evaluate their utility for assessing painful responses in this population. The study will be a 2-week, open-label study conducted at a single study site in patients with pain associated with patellar tendinopathy in a single knee. During this out-patient study, patients will apply one study patch to the affected tendon twice daily for approximately 14 days. Patches will be applied morning and evening (applications separated by approximately 8-10 hours) and removed after 2-4 hours.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* have pain associated with patellar tendinopathy in a single knee (minimum 2-week duration)
* have tenderness at the proximal insertion of the patellar tendon in the affected knee

Exclusion Criteria:

* have any history of surgery in the target knee
* have used any topically applied pain medication on the target treatment area within 3 days preceding the Screening/Baseline Visit
* have had any injected steroids in the target knee within 3 months of the Screening/Baseline Visit
* have used any injected pain medication within 14 days preceding the Screening/Baseline Visit
* are receiving class 1 antiarrhythmic drugs (ie, tocainide, mexiletine, etc.)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment (VISA) score | Two weeks
  VISA questionnaire, an index of severity and symptoms of patellar tendinopathy, completed by the patient (beginning and end of the study).

SECONDARY OUTCOMES:
Pain intensity | Two weeks
Patient Global Assessment of Treatment Satisfaction (PGAS) | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henry Goitz, MD, Principal Investigator — Detroit Medical Center, Sports Medicine Clinic
Locations (1):
- Sports Medicine Clinic, Warren, Michigan, United States